CLINICAL TRIAL: NCT04924647
Title: Lenalidomide and Dexamethasone for Rosai-Dorfman Disease: A Single Arm, Single Center, Prospective Phase 2 Study
Brief Title: Lenalidomide and Dexamethasone for Rosai-Dorfman Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Cao Xinxin, Associate Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHRDD1
Record Dates: First submitted 2021-06-07; First posted 2021-06-14 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Rosai-Dorfman Disease
Keywords: Rosai-Dorfman Disease; lenalidomide; dexamethasone
MeSH Terms: conditions — Histiocytosis, Sinus | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RD (Experimental): lenalidomide and dexamethasone
  Interventions: Drug: lenalidomide and dexamethasone

INTERVENTIONS:
Drug: lenalidomide and dexamethasone — lenalidomide 25mg d1-21 and dexamethasone 20-40mg d1，8，15，22

SUMMARY:
Rosai-Dorfman Disease (RDD) is a rare, heterogeneous histiocytic disorder. Because of the rarity of RDD and a lack of prospective randomized trials, the treatment strategy for RDD is mostly based on retrospective study. Steroid was suggested as frontline treatment as RDD with only lymph nodes involvement. Studies showed thalidomide or lenalidomide showed some effect in recurrent/refractory skin RDD. The investigators want to analyze the efficacy and toxicity of lenalidomide combined with dexamethasone regimens in the treatment of RDD among adult patients at our hospital.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of RDD
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
* Patients must have adequate renal, liver, and bone marrow function as defined by the following criteria:

Absolute neutrophil count ≥1500 cells per mm3 Platelet count ≥100000 cells per mm3 Creatinine clearance [according to Cockcroft formula] ≥60 mL/min. Aspartate aminotransferase and alanine aminotransferase ≤2·5×upper limit of normal [ULN], and total bilirubin ≤2·5×ULN; or ≤10×ULN in the case of known liver involvement by RDD.

* No active or untreated infection.
* No cardiac abnormalities.
* Subject provide written informed consent.
* A female is eligible to enter and participate in this study if she is of:

Non-childbearing potential including ω Any female who has had a surgical procedure rendering her incapable of becoming pregnant.

ω Subjects have experienced total cessation of menses for more than 1 year and be greater than 45 years in age.

⎫ Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, and agrees to use adequate contraception.

• Male subjects must use an effective barrier method of contraception during the study and for 90 days following the last course of MA if sexually active with a childbearing potential

Exclusion Criteria:

* Patients had concurrent malignancies.
* History of myocardial infarction, or unstable angina, or New York Heart Association (NYHA) Grade III-IV within 6 months prior to Day 1.
* Women who were pregnant or of childbearing potential.
* Known HIV seropositive, active hepatitis C infection, and/or hepatitis B (defined as HCV RNA≥1000 copies or HBV DNA ≥1000 copies at screening).
* Major surgical procedure within 28 days prior to the first dose of study treatment.
* Presence of uncontrolled infection.
* Evidence of active bleeding or bleeding diathesis.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Event-free survival | the duration from initiation of treatment to the date of first documented event or date of death from any cause, whichever come first, assessed up to 5 years
  Events were defined as a poor response to RD, reactivation after RD therapy and death from any cause.

SECONDARY OUTCOMES:
Overall response rate | on 12 months
  the cumulative number of patients with either non-active disease or regressive disease (signs and symptoms were improved with no new lesions) after RD
Overall survival | the duration from initiation of RD treatment to the date of death or last follow-up, assessed up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dao-bin Zhou, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

REFERENCES:
- [Derived] Chang L, Lang M, Liu T, Lin H, Liu ZZ, Cai H, Zhou DB, Cao XX. Lenalidomide and dexamethasone for Rosai-Dorfman disease: a single arm, single center, prospective phase 2 study. EClinicalMedicine. 2024 Jun 21;73:102685. doi: 10.1016/j.eclinm.2024.102685. eCollection 2024 Jul. PMID 39022796